CLINICAL TRIAL: NCT01359033
Title: Compare the Patient Risk and Between-hospital Variation in Myocardial Infarction Mortality in the United Kingdom and Sweden
Brief Title: MI Mortality Risk and Between-hospital Risk Variation in the United Kingdom and Sweden
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: NICOR/MINAP, the United Kingdom (Unknown); National Institute for Cardiovascular Outcomes Research (Other); MINAP: Myocardial Ischaemia National Audit Project (Unknown); SWEDEHEART/RIKS-HIA, Sweden (Unknown); SWEDEHEART: Swedish Web-System for Enhancement and Development of Evidence-Based Care in Heart Disease Evaluated According to Recommended Therapies (Unknown); RIKS-HIA: Register of Information and Knowledge about Swedish Heart Intensive care Admissions (Unknown)
Responsible Party: Sponsor
Other Study IDs: FP7-EIS-WP7-MINAP
Record Dates: First submitted 2011-05-23; First posted 2011-05-24 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2014-02

CONDITIONS: Acute Myocardial Infarction
Keywords: Myocardial Infarction; UK; Sweden; National audit registry; MINAP; RIKS-HIA
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MINAP cohort: The Myocardial Ischaemia National Audit Project (MINAP) was established in 1999, in response to the national service framework (NSF) for coronary heart disease, to examine the quality of management of heart attacks (myocardial infarction) in hospitals in England and Wales.
- RIKS-HIA cohort: The Register of Information and Knowledge About Swedish Heart Intensive Care Admissions (RIKS-HIA) has been established to record clinical and treatment information for all patients admitted to the coronary care units in Sweden from 1995.

SUMMARY:
The study aims to investigate the differences in survival trajectories and hospital variability in myocardial infarction (MI) mortality rates in the UK and Sweden.

DETAILED DESCRIPTION:
Limited evidence is available in comparing hospital level care and reference mortality risks between countries, due to the scarce availability of nationwide coronary heart disease data. The demographics and medical expenditure percentage are comparable in the United Kingdom and Sweden; however, the in-hospital case-fatality rates within 30 days after admission for acute myocardial infarction was greater in the UK than Sweden (6.3% versus 2.9%)(OECD, 2009). To investigate the discrepancy, the current study aims to compare the mortality risk differences and associated explanatory factors between the two countries. Results of the study can contribute to myocardial infarction care implementation in the UK and Sweden.

The UK Myocardial Ischaemia National Audit Project (MINAP)and Register of Information and Knowledge about Swedish Heart Intensive care Admissions (RIKS-HIA) are few quality national registries currently available for acute coronary syndrome. Using data from the MINAP and RIKS-HIA, we propose to investigate (1)the survival trajectories for a reference patient with myocardial infarction and (2) hospital variability in myocardial infarction mortality rate in the UK and Sweden, adjusted for important patient-level and hospital-level covariates.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 30 years old who had hospital admission for acute myocardial infarction.
* Admission period ranged from 1st January, 2004 to 31th December, 2008.

Exclusion Criteria:

* Patients with missing data in the admission time and/or primary outcomes.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the UK, all patients with an admission recorded in the MINAP database during 1st January 2004 and 31 December 2008 in 253 hospitals in England and Wales will be included in the study. For Sweden, all patients with an admission recorded in the RIKS-HIA during 1st January 2004 and 31 December 2008 in 74 hospitals in Sweden will be included. Only patients with acute myocardial infarction will be included as the study population.
Sampling Method: Non-Probability Sample
Enrollment: 510863 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30-day
  all-cause mortality at 30-day following hospitalization for acute Myocardial Infarction

SECONDARY OUTCOMES:
1-year mortality | 1 year
  all-cause mortality at 1-year following hospitalization for acute Myocardial Infarction

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Chia Chung, Ph.D, Principal Investigator — University College, London
Locations (2):
- Uppsala Clinial Research Center, Uppsala, Sweden
- University College London, London, United Kingdom

REFERENCES:
- [Background] Rosvall M, Ohlsson H, Hansen O, Chaix B, Merlo J. Auditing patient registration in the Swedish quality register for acute coronary syndrome. Scand J Public Health. 2010 Jul;38(5):533-40. doi: 10.1177/1403494810365109. Epub 2010 Apr 20. PMID 20406796
- [Background] Jernberg T, Attebring MF, Hambraeus K, Ivert T, James S, Jeppsson A, Lagerqvist B, Lindahl B, Stenestrand U, Wallentin L. The Swedish Web-system for enhancement and development of evidence-based care in heart disease evaluated according to recommended therapies (SWEDEHEART). Heart. 2010 Oct;96(20):1617-21. doi: 10.1136/hrt.2010.198804. Epub 2010 Aug 27. PMID 20801780
- [Background] Birkhead JS, Walker L, Pearson M, Weston C, Cunningham AD, Rickards AF; National Audit of Myocardial Infarction Project Steering Group. Improving care for patients with acute coronary syndromes: initial results from the National Audit of Myocardial Infarction Project (MINAP). Heart. 2004 Sep;90(9):1004-9. doi: 10.1136/hrt.2004.034470. PMID 15310686
- [Background] Birkhead JS, Weston C, Lowe D. Impact of specialty of admitting physician and type of hospital on care and outcome for myocardial infarction in England and Wales during 2004-5: observational study. BMJ. 2006 Jun 3;332(7553):1306-11. doi: 10.1136/bmj.38849.440914.AE. Epub 2006 May 16. PMID 16705004
- [Derived] Chung SC, Sundstrom J, Gale CP, James S, Deanfield J, Wallentin L, Timmis A, Jernberg T, Hemingway H; Swedish Web-System for Enhancement and Development of Evidence-Based Care in Heart Disease Evaluated According to Recommended Therapies/Register of Information and Knowledge about Swedish Heart Intensive care Admissions; National Institute for Cardiovascular Outcomes Research/Myocardial Ischaemia National Audit Project; CAardiovascular Disease Research Using Linked Bespoke Studies and Electronic Health Records. Comparison of hospital variation in acute myocardial infarction care and outcome between Sweden and United Kingdom: population based cohort study using nationwide clinical registries. BMJ. 2015 Aug 7;351:h3913. doi: 10.1136/bmj.h3913. PMID 26254445
- [Derived] Chung SC, Gedeborg R, Nicholas O, James S, Jeppsson A, Wolfe C, Heuschmann P, Wallentin L, Deanfield J, Timmis A, Jernberg T, Hemingway H. Acute myocardial infarction: a comparison of short-term survival in national outcome registries in Sweden and the UK. Lancet. 2014 Apr 12;383(9925):1305-1312. doi: 10.1016/S0140-6736(13)62070-X. Epub 2014 Jan 23. PMID 24461715
- See also: Myocardial Ischaemia National Audit Project (MINAP) — http://www.hqip.org.uk/myocardial-ischaemia-national-audit-project-minap/
- See also: The Register of Information and Knowledge about Swedish Heart Intensive care Admissions — http://www.ucr.uu.se/rikshia/